CLINICAL TRIAL: NCT01498588
Title: Phase II Neoadjuvant Trial of Eribulin Followed by Dose Dense Doxorubicin and Cyclophosphamide for Her2-negative, Locally Advanced Breast Cancer
Brief Title: Trial of Eribulin Followed by Doxorubicin & Cyclophosphamide for Her2-negative, Locally Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Keerthi Gogineni, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00050068; WCI1937-10 (Other: Other)
Record Dates: First submitted 2011-10-13; First posted 2011-12-23 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasms; Breast Cancer; Breast Tumors; Cancer of the Breast; Neoplasms, Breast; Tumors, Breast
Keywords: Breast Neoplasms; Breast Cancer; Breast Tumors; Cancer of the Breast; Neoplasms, Breast; Tumors, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Doxorubicin; Cyclophosphamide; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eribulin+Doxorubicin+Cyclophosphamide (Experimental): Neoadjuvant eribulin followed by dose-dense doxorubicin and cyclophosphamide
  Eribulin Day 1 and Day 8 of a 21 day cycle x 4 cycles:
  Day 1: Eribulin 1.4mg/m² IV
  Day 8: Eribulin 1.4mg/m² IV
  Dose-dense doxorubicin and cyclophosphamide every 14 days x 4 cycles:
  Day 1: Doxorubicin 60mg/m² IV
  Day 1: Cyclophosphamide 600mg/m² IV
  Day 2: Pegfilgrastim support 6mg sc at least 24 hours after chemotherapy at the discretion of the investigator.
  Interventions: Drug: Eribulin; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Eribulin — Patients will receive 4 cycles of neoadjuvant eribulin followed by 4 cycles of dose-dense doxorubicin and cyclophosphamide (AC).
  Other Names: Halaven
Drug: Doxorubicin — Neoadjuvant eribulin followed by dose-dense doxorubicin and cyclophosphamide
  Other Names: Adriamycin
Drug: Cyclophosphamide — Neoadjuvant eribulin followed by dose-dense doxorubicin and cyclophosphamide
  Other Names: Cytoxan
Drug: Pegfilgrastim — Growth factor support (pegfilgrastim) can be given at the discretion of the investigator. Administration of pegfilgrastim is required 24 to 48 hours following administration of dose-dense doxorubicin and cyclophosphamide.
  Other Names: Neulasta

SUMMARY:
Previous studies have shown that chemotherapy has the same effect on treating breast cancer whether you receive it before or after surgery. Receiving chemotherapy before surgery, rather than after surgery, may allow the patient to have less extensive surgery. The purpose of this study is to identify new treatment regimens with better response rates and to find out if the combination of eribulin followed by doxorubicin and cyclophosphamide can shrink the size of the patient's breast tumor and allow you to preserve your breast. Additionally, by receiving chemotherapy before surgery, the investigators will be able to determine if your cancer is responsive to chemotherapy.

DETAILED DESCRIPTION:
This is a phase 2, single-arm, open label study. Patients with Her2-negative, locally advanced breast cancer will be enrolled on the study prior to receiving neoadjuvant chemotherapy. Patients will receive 4 cycles of neoadjuvant eribulin followed by 4 cycles of dose-dense doxorubicin and cyclophosphamide (AC).

All patients will have a baseline biopsy prior to study entry to determine eligibility. Patients will undergo repeat breast imaging and optional biopsy after completing 4 cycles of eribulin. Patients will then receive 4 cycles of dose-dense AC. Patients will undergo repeat breast imaging followed by surgical resection within 30 days of completing last cycle of chemotherapy. Patients who are not surgical candidates after completion of chemotherapy will be asked to undergo optional repeat biopsy prior to receiving additional treatment at the discretion of the investigator. Patients will continue to be followed per standard practice guideline after surgery

Clinical response will be determined by clinical breast examination prior to each cycle of chemotherapy and by breast imaging performed at baseline, after completion of eribulin, and prior to surgery. Pathologic complete response (pCR) will be determined at the time of surgical resection. Correlative biomarker studies will be performed on tumor samples at the completion of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast carcinoma.
* Locally advanced breast cancer (Stage IIIA to IIIC).
* Invasive breast cancer must be Her2-negative. If breast cancer is Her2 2+ by immunohistochemistry (IHC), then fluorescence in situ hybridization (FISH) must be negative for Her2 gene amplification.
* No evidence of disease outside the breast or chest wall, except ipsilateral axillary lymph nodes on staging scans (CT chest/abdomen/pelvis and bone scan or positron emission tomography [PET] scan).
* Patients must have measurable disease as defined by palpable lesion with both diameters ≥ 1 cm measurable with caliper and/or a positive mammogram or ultrasound with at least one dimension ≥ 1 cm. Bilateral mammogram and clip placement is required for study entry. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within the 14 days if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a mammogram or MRI must be done within 2 months prior to study entry. If clinically indicated, xrays and scans must be done within 28 days of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 within 14 days of study entry.
* Normal (greater than 50%) left ventricular ejection fraction (LVEF) by multigated acquisition (MUGA) scan or echocardiography.
* Signed informed consent.
* Adequate organ function within 2 weeks of study entry:

  * Absolute neutrophil count ≥ 1500/mm³, Hgb ≥ 9.0 g/dl and platelet count ≥ 100,000/mm³.
  * Total bilirubin ≤ upper limit of normal.
  * Creatinine ≤ 1.5 mg/dL or calculated creatinine clearance rate (CrCL) ≥ 50 mL/min using the Cockroft Gault equation.
  * Serum glutamate oxaloacetate transaminase (SGOT)/(AST) or serum glutamate pyruvate transaminase (SGPT)/(ALT) and alkaline phosphatase (alk phos) must be within the range allowing for eligibility.
* Patients must be over 18 years old.
* International normalized ratio (INR) < 1.5 or a prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation.
* Patient must have signed informed consent prior to registration on this study.

Exclusion Criteria:

* Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer. Patients with history of breast cancer greater than 5 years from initial diagnosis are eligible for the study. Patients may not have received anthracycline-based chemotherapy in the past. Patients with history of ductal carcinoma in situ (DCIS) are eligible if there were treated with surgery alone.
* Medical, psychological or surgical condition which the investigator feels might compromise study participation.
* History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible.
* Evidence of sensory and/or peripheral neuropathy > grade 1.
* Serious, uncontrolled, concurrent infection(s).
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Pregnant or lactating women are not eligible. Women of childbearing potential must have a negative serum or urine pregnancy test completed within 7 days of study treatment. Women or men of childbearing potential not using a reliable and appropriate contraceptive method are not eligible. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Thromboembolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Cardiac disease: congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keerthi Gogineni, MD, MSHP, Principal Investigator — Emory University Winship Cancer Institute
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to accrual from October 2011 to June 2015. Enrolled participants were from Winship Cancer Institute of Emory University and Emory University Hospital Midtown.
Groups:
- Eribulin+Doxorubicin+Cyclophosphamide: Neoadjuvant eribulin followed by dose-dense doxorubicin and cyclophosphamide
  Eribulin Day 1 and Day 8 of a 21 day cycle x 4 cycles:
  Day 1: Eribulin 1.4mg/m² IV
  Day 8: Eribulin 1.4mg/m² IV
  Dose-dense doxorubicin and cyclophosphamide every 14 days x 4 cycles:
  Day 1: Doxorubicin 60mg/m² IV
  Day 1: Cyclophosphamide 600mg/m² IV
  Day 2: Pegfilgrastim support 6mg sc at least 24 hours after chemotherapy
Period: Overall Study
Arm/Group | Eribulin+Doxorubicin+Cyclophosphamide
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eribulin+Doxorubicin+Cyclophosphamide
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate at the Time of Surgery
Description: Patients will receive treatment for 20 weeks with primary outcome measured at the time of surgery. Surgery is typically 4-6 weeks after completion of chemotherapy, so patients will be on study for 24 weeks on average. Response was measured by pathologist's standard of care assessment of extent of residual disease. If the patient had no evidence of invasive or in situ residual disease present in the breast and lymph node (i.e. ypT0N0), then this was defined as a pathologic complete response (pCR). Reported is the number of participants showing pCR.
Time Frame: Average of 24 weeks
Population: Pathology information at the time of definitive resection was available for six of seven patients. One patient was ultimately lost to follow-up.
Measure: Number; unit: participants
Arm/Group | Eribulin+Doxorubicin+Cyclophosphamide
Number analyzed (Participants) | 7
participants
  Pathologic Complete Response (pCR) | 1
  No pCR | 5
  Unknown | 1

2. Secondary Outcome: Toxicity of Chemotherapy Regimen (Number of Participants With Any Adverse Events)
Description: Toxicity of chemotherapy at each physician visit using Common Toxicity Criteria for Adverse Effects (CTCAE) criteria.
Time Frame: Through 20 weeks of chemotherapy
Measure: Number; unit: participants
Arm/Group | Eribulin+Doxorubicin+Cyclophosphamide
Number analyzed (Participants) | 7
participants | 2

ADVERSE EVENTS:
Arm/Group | Eribulin+Doxorubicin+Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin+Doxorubicin+Cyclophosphamide (N=7)
Fatigue (General disorders) | 1
Insomnia (General disorders) | 1
Neuropathy (Nervous system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Hemorrhage (Blood and lymphatic system disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Elevated ALT (Metabolism and nutrition disorders) | 1
Elevated AST (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Study accrual was low at 7 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes